CLINICAL TRIAL: NCT04796298
Title: Effect of Ballistic Stretching, Extender Exercise, and Kinesio Taping on Hamstring Viscoelasticity and Rower Athletic Performance - A Preliminary Study
Brief Title: Interventions and Viscoelasticity of Hamstring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Principal Investigator, Onur Atakan Sekibağ, Physiotherapist, Yeditepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASekibag
Record Dates: First submitted 2021-03-07; First posted 2021-03-12 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Injury; Back, Lower, Superficial; Hamstring Injury; Sport Injury; Sports Physical Therapy
Keywords: Ballistic Stretching; Eccentric exercise; Kinesiotaping; Viscoelasticity; Hamstrings; Athletic Performance; Rowers
MeSH Terms: conditions — Wounds and Injuries | interventions — Athletic Tape

STUDY DESIGN:
Intervention Model Description: Study is designed as Randomized Uncontrolled Trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ballistic Hamstring Stretching Group (Experimental): Ballistic Hamstring Stretching
  Interventions: Procedure: Ballistic Hamstring Stretching
- Hamstring Extender Exercise Group (Experimental): Hamstring Extender Exercise
  Interventions: Procedure: Hamstring Extender Exercise
- Kinesiotape Group (Experimental): Kinesiotape
  Interventions: Procedure: Kinesiotape

INTERVENTIONS:
Procedure: Ballistic Hamstring Stretching — Athletes were asked to reach the floor in the BS group by leaning over in the standing posture without knee flexion. When they feel the tension in hamstring muscle groups, athletes were requested to make small rebounding motion at degrees between 3°-5° for half a minute.
  Arms: Ballistic Hamstring Stretching Group
Procedure: Hamstring Extender Exercise — Athletes were asked to applied 12 repetitions and 3 sets of hamstring extender exercise. Firstly athlete lies on his/her back. Then, athlete is asked to do 90 degrees of knee and hip flexion at the same time. Finally, the person is expected to perform slow repetitive knee extension to the point of maximal possible extension.
  Arms: Hamstring Extender Exercise Group
Procedure: Kinesiotape — Kinesio tape is applied on the hamstring muscle with a Y shape and %25 tension force.
  Arms: Kinesiotape Group

SUMMARY:
The study aims to investigate acute effects of ballistic hamstring stretching, hamstring extender exercise, and kinesiotaping application on viscoelasticity of hamstrings and standing long jump performance on rowers.

DETAILED DESCRIPTION:
The study aims to investigate acute effects of ballistic hamstring stretching, hamstring extender exercise, and kinesiotaping application on viscoelasticity of hamstrings and standing long jump performance on rowers. A total of 60 professional rowing athletes were included. Viscoelasticity of hamstrings were assessed by MyotonPRO, Tallinn, Estonia. Athletic performance was assessed by Standing Long Jump Test (SLJT). The athletes were randomly divided into Ballistic Hamstring Stretching Group (n= 20), Hamstring Extender Exercise Group (n= 20), and Kinesiotape Group (n= 20). For balistic hamstring stretching, athletes were asked to reach the floor in the BS group by leaning over in the standing posture without knee flexion. When they feel the tension in hamstring muscle groups, athletes were requested to make small rebounding motion at degrees between 3°-5° for half a minute. For hamstring extender exercise, athletes were asked to apply the exercise 12 repetitions and 3 sets. Kinesiotaping was applied on the hamstring muscle with Y shape and 25% tension force.

ELIGIBILITY:
Inclusion Criteria:

* Participating to the study in a voluntary basis.
* Athletes with 14-18 years old.
* Being a rowing athlete for at least a year.
* Being an athlete in Fenerbahce Rowing Team and Turkish Divers Club - Rowing Branch.

Exclusion Criteria:

* Having a musculoskeletal injury involving the lower extremity in the last 6 months.
* Having undergone a surgical operation in the last 6 months.
* Any limitation in lower extremity range of motion.
* Failing to complete the Ballistic Hamstring Stretching, Hamstring Extender Exercise or Kinesio taping Application.
* Wanting to quit from study.

Ages: 14 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Frequency of Muscle (F) | Day 1
  The tones of muscle is described by frequency of muscle or oscillation frequency (Hz). It is examined by the MyotonPro, Tallinn, Estonia.
Stiffness of Muscle (S) | Day 1
  Stiffness of Muscle is described by reaction to contraction or forces from outside of tissue that may cause the original form to deteriorate. It is examined by the MyotonPro, Tallinn, Estonia.
Decrement of Muscle (D) | Day 1
  The elasticity of a muscle is described by a logarithmic reduction of tissue's normal amplitude. It is more related with the dissipation of mechanical energy that arises between the deformation of the tissue and its recovery. It is a biomechanical feature of tissue that is called as elasticity. It is examined by the MyotonPro, Tallinn, Estonia.
Relaxation of Muscle (R) | Day 1
  It is the time which is called as Mechanical Stress Relaxation Time (ms) between the deformation of the normal shape of the tissue and its return to its original shape. It is examined by the MyotonPro, Tallinn, Estonia.
Creep of Muscle (C) | Day 1
  It is defined as ratio of deterioration and relaxation time of tissue. In case of a continuous stress, tissue regularly stretches over time. This is called as creep. It is examined by the MyotonPro, Tallinn, Estonia.
Athletic Performance | Day 1
  Athletic Performance is assessed by Standing Long Jump Test. It is a horizontal jump test that measures anaerobic performance.

CONTACTS AND LOCATIONS:
Overall Officials: Onur Atakan Sekibağ, MSc, Principal Investigator — Yeditepe University, Health Sciences Faculty, Department of Physiotherapy and Rehabilitation; Şule Badıllı Demirbaş, Asst. Prof., Study Chair — Yeditepe University, Health Sciences Faculty, Department of Physiotherapy and Rehabilitation; Ayça Yağcıoğlu, MSc, Study Chair — Yeditepe University, Health Sciences Faculty, Department of Physiotherapy and Rehabilitation
Locations (1):
- Yeditepe University, Health Sciences Faculty, Department of Physiotherapy and Rehabilitation, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No